CLINICAL TRIAL: NCT03822247
Title: A Prospective, Randomized Comparison of Multidisciplinary Recovery After Surgery Program and Conventional Protocol for Perioperative Care in Orthopedics and Traumatology
Brief Title: Evaluation of Multidisciplinary Recovery After Surgery Program in Orthopedics and Traumatology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Klinički Bolnički Centar Zagreb (Other)
Responsible Party: Principal Investigator, Nikica Darabos, Assistant Professor, Klinički Bolnički Centar Zagreb
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KBC Zagreb Surgery
Record Dates: First submitted 2019-01-27; First posted 2019-01-30 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Hip Fractures; Knee Fracture; Hip Arthritis; Knee Arthritis
Keywords: Recovery; Patient reported outcome measures; Hip fracture; Hip arthritis; Knee fracture; Knee arthritis
MeSH Terms: conditions — Hip Fractures; Knee Fractures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multidisciplinary Recovery Program (Experimental): Two cohorts of patients will randomly be placed in either experimental od no intervention group.
  Patients undergoing Multidisciplinary Recovery After Surgery Program will gain better preparation for early mobilization after surgery, nutritional support, individually modified analgesia and psychological support during inpatient treatment. Program includes preoperative, intraoperative and postoperative multidisciplinary comprehensive interventions.
  Interventions: Procedure: Multidisciplinary Recovery Program
- Conventional Perioperative Care (No Intervention): Patients undergoing conventional care

INTERVENTIONS:
Procedure: Multidisciplinary Recovery Program — Preoperative care:
  * Patient's education
  * Providing respiratory training
  * Assessment of nutritional status
  * Application of compression stockings
  * Thromboembolism prophylaxis by low molecular weighted heparin
  * Induction of hemodynamic support 12 hours before the surgery
  * Oral carbohydrate solution loading until 2 hours before the surgery
  Intraoperative care:
  * Maintaining normothermia
  * Multimodal prevention of postoperative nausea and vomiting
  * Use of spinal anesthesia
  * Prevention of excessive blood loss
  * Local anesthetic infiltration
  Postoperative care:
  * Active pain control
  * Early mobilization
  * Early onset of oral nutrition
  * Early delirium detection
  * Application of compression stockings
  Arms: Multidisciplinary Recovery Program

SUMMARY:
The aim of the recovery protocol is to reduce surgical trauma, postoperative pain, and complications, shorten hospital treatment and improve postoperative recovery. Orthopedic and traumatology surgeries are often followed by a long-lasting recovery with difficulties of everyday functioning. Up to this time, only a few publications of multidisciplinary protocol in orthopedics and traumatology have been published, mostly to improve the care of patients after elective surgical procedures. The goal of multidisciplinary after surgery recovery program in orthopedics and traumatology is to improve the care of both urgent and elective patients using standardized, multi-professional care programs. It focuses on patient education, preoperative respiratory training, adequate nutritive and hemodynamic support, modified anesthesia protocol, prevention of postoperative pain, nausea and vomiting, and early postoperative delirium detection. The implementation of the program will reduce the rate of postoperative complications and the rate of rehospitalization, enhance the recovery after surgery and increase the satisfaction with the treatment.

DETAILED DESCRIPTION:
The protocol combines scientifically proven interventions to standardize medical care, improve treatment outcomes and reduce healthcare costs. The aim is to reduce surgical trauma and postoperative pain, reduce complications, shorten hospital treatment and improve postoperative recovery. Moreover, it has been shown that using standardized, patient oriented recovery protocol significantly improves the outcomes and quality of care, but also brings financial benefit for the hospital as well as for the health system in general. Studies about implementing multidisciplinary recovery protocol in orthopedic and traumatology are scarce. Orthopedic and traumatology surgeries are often followed by a long-lasting and demanding recovery characterized by the difficulties of everyday functioning. Recovery is therefore multidisciplinary: for example, it is necessary to monitor the nutritional status of a patient, decrease postoperative pain, monitor cognitive status, etc. Until now only a few publications of recovery protocols in orthopedics and traumatology have been published, mostly to improve the care of patients after elective surgical procedures. The goal of this protocol in orthopedics and traumatology is to improve the care of both urgent and elective patients using standardized, multi-professional care programs. It was created based on evidence-based practice and modified by multidisciplinary team of orthopedic and traumatology surgeons, anesthesiologists, physiatrist, physiotherapists, specialized medical nurses, nutritionists, and psychiatrists. It focuses on patient preoperative education, preoperative respiratory training, adequate nutritive and hemodynamic support, modified local and regional anesthesia protocol, prevention of postoperative pain, nausea and vomiting, and early postoperative delirium detection. The investigators postulate that the implementation of this program will reduce the rate of postoperative complications and the rate of rehospitalization, enhance the recovery after surgery and increase the satisfaction with the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Fracture od proximal femur or knee fracture requiring surgery
* Hip or knee arthrosis requiring joint replacement
* American Society of Anesthesiologists (ASA) score II or III
* Ability to provide informed consent

Exclusion Criteria:

* Severe cognitive impairment
* Pregnancy
* End stage of malignant disease
* Decompensated heart or liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-08-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Early Postoperative Complications | 48 hours after surgery
  Occurrence of early complications:
  * Dislocation or malpositioning of joint replacement
  * Neurological deficit
  * Need for blood transfusion
  * Postoperative delirium
  * Nausea or vomiting
  * Pneumonia
  * Headache
  * Wound dehiscence, secretion, inflammation, bleeding
Late Postoperative Complications | 10 days after surgery
  Occurrence of late complications:
  * Wound infection, healing by secundam
  * Decubitus
  * Fracture of joint replacement
  * Aseptic loosening of hip joint replacement
  * Infection of joint replacement
  * Thromboembolism
  * Need for a revision

SECONDARY OUTCOMES:
Readmission rates | 30 days after surgery
  Rate of readmission to the hospital
Patient-reported outcome after orthopedic surgery using The Western Ontario and McMaster Universities Arthritis Index (WOMAC) | 2 days, 60 days after surgery, 90 days after surgery
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is a self-administered questionnaire consisting of 24 items divided into 3 subscales (pain, stiffness and physical function). The questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. A sum of the scores for all three subscales gives a total WOMAC score; higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Pain assessment using Visual Analog Scale (VAS) | 1 day, 2 days, 60 days after surgery, 90 days after surgery
  The Visual Analog Scale (VAS) is a unidimensional measure of pain intensity. It is a straight horizontal line of fixed length of 100 mm. The ends are defined as the extreme limits of pain orientated from the left (worst) to the right (best). The score represents the distance measured (mm) between the worst and best mark, providing a range of scores between 0-100. A higher score indicates greater pain intensity. The following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm).
Assessment of health related quality of life using Euro Quality of Life Index (Euro QoL 5-D 5-L) | baseline, 2 days, 60 days after surgery, 90 days after surgery
  The instrument Euro Quality of Life Index (Euro QoL 5-D 5-L) measures five dimensions, Mobility, Self-care, Daily activities, Pain/Discomfort, Anxiety/ Depression. Each dimension can be rated at five levels: from no problems to major problems. The five dimensions can be summed into a descriptive health state with 11111 representing no problems in any of the five health dimensions and 55555 indicating major problems in any of the five health dimensions. Second part of the instrument is the Visual Analogue Scale to assess health status at baseline, where 0 signifies worst imaginable health state, and 100 signifies best imaginable health state.
Evaluation of patients' satisfaction with the care provided using The Short-form patient satisfaction questionnaire (PSQ-18) | 3 days after surgery
  The Short-form patient satisfaction questionnaire (PSQ-18) contains 18 items tapping each of the seven dimension of satisfaction with medical care: general satisfaction, technical quality, interpersonal manner, communication, financial aspects, time spent with the doctor and accessibility and convenience. All items are scored so that high scores reflect satisfaction with medical care and after item scoring, items within the same subscale should be averaged together to create the seven subscale scores.

CONTACTS AND LOCATIONS:
Overall Officials: Nikica Daraboš, Study Chair — Head of Department of traumatology, bone and joint surgery
Locations (1):
- KBC Zagreb, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No